CLINICAL TRIAL: NCT06983548
Title: Chikungunya Virus Detection in Semen: Preliminary Study - CHIKSPERM
Brief Title: Chikungunya Virus Detection in Semen
Acronym: CHIKSPERM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Agence de La Biomédecine (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/25/0186; 2025-A00823-46 (Other: ANSM)
Record Dates: First submitted 2025-04-15; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Chikungunya Virus Infection
Keywords: Chikungunya; semen analysis; viral excretion; RT-PCR
MeSH Terms: conditions — Chikungunya Fever | interventions — Seeds; Blood Specimen Collection; Urinalysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chikungunya virus-infected men (Other)
  Interventions: Biological: semen, blood and urine tests

INTERVENTIONS:
Biological: semen, blood and urine tests — Patients will undergo several tests, including semen analysis, spermocytogram, blood and urine tests, serology, and RT-PCR. These tests will be conducted on days 7±2, 15±2, 30±3, 60±5, 90±5, and 180±15. (Patients will only undergo the V6 if the sperm PCR result comes back positive on D90).

SUMMARY:
Chikungunya is an arboviral disease transmitted by Aedes mosquitoes, present in intertropical zones and Europe. In August 2024, autochthonous cases appeared on Réunion, followed by a large epidemic. In March 2025, the incidence surpassed 2,000 cases per week. Due to a lack of data, the Haut Comité de Santé Publique issued an unfavorable opinion on using substances of human origin during the epidemic.

Although the presence of Chikungunya virus genome in semen has been reported in 7 men, the incidence of viral excretion is unknown. This raises concerns about the risk of sexual transmission and infectivity, especially in assisted reproductive technologies. Previous studies on other arboviruses (Zika, dengue) have explored genital excretion.

The goal of this prospective pilot study is to investigate Chikungunya virus presence and infectivity in semen, as well as to evaluate the effectiveness of sperm preparation methods in obtaining virus-free gametes. Fifteen patients with acute Chikungunya virus infection will provide blood, urine, and semen samples at different time points (7, 15, 30, 60, 90, and 180 days post-symptom onset). Seminal plasma, native sperm cells, and prepared sperm fractions will be tested for Chikungunya virus RNA at the University Hospital of La Réunion and Toulouse.

This study will provide insights into viral excretion patterns and help improve the safety of medically assisted reproduction in epidemic situations.

DETAILED DESCRIPTION:
Chikungunya is an arbovirosis transmitted by mosquitoes of the genus Aedes. These vectors are present in intertropical zones, but have also been present in Europe for several years. The chikungunya virus (CHIKV) is a virus of the Alphavirus genus and the Togaviridae family. In mid-August 2024, autochthonous cases of chikungunya appeared on Réunion, followed by a vast epidemic, leading to the activation of a level 3 ORSEC plan, then level 4 in March 2025. At this time, the incidence was over 2,000 cases per week. In the absence of data, and as a precaution, the Haut Comité de Santé Publique issued an unfavourable opinion on the use of substances of human origin during the 2025 epidemic. Epidemics seem to recur in intertropical zones and could emerge in mainland France due to the presence of a vector (Ae. albopictus).

At present, only two case studies have reported the presence of the CHIKV genome in the semen of 7 men, but the incidence of positive semen in infected men is unknown. This genital excretion has already been described for other arboviruses belonging to the Flaviviridae family, such as Zika fever and dengue fever.

The possibility of detecting the CHIKV genome in semen raises questions about its frequency and kinetics, the infectivity of the virus and the risk of sexual transmission of the virus or during assisted reproductive technologies. It is therefore essential to: 1) understand the kinetics of viral excretion in semen and urine compared with the viremia used to diagnose infection, 2) study the fractions of semen containing viral genomes and 3) investigate possible infectivity (seminal plasma, native sperm cells, spermatozoa). We benefit from the experience of pilot studies carried out under the same conditions on other viruses (HIV, HCV, ZIKV, DENV SARS-CoV-2).

The aim of this project, carried out within teams involved in the virus and reproduction theme, is to investigate the presence of the CHIKUNGUNYA virus in sperm (genome and infectivity), to specify its location, and to study the effectiveness of conventional sperm preparation methods in obtaining virus-free gametes.

This is a prospective, pilot study involving 15 patients in the acute phase of infection with positive CHIKV RNA detection in blood and/or urine. Blood, urine and semen samples will be taken 7 days after the onset of clinical signs and 15, 30, 60, 90 and 180 days later.

In the genital compartment, CHIKV RNA will be tested in seminal plasma, in native sperm cells and in cell fractions obtained after sperm preparation. The semen will be processed at the Reproduction Centre of the University Hospital of La Réunion, and the CHIKV RNA will be tested in the different aliquots in the virology laboratory of the University Hospital of Toulouse.

This study will make it possible to determine the frequency of viral excretion in the semen and to determine how this changes during the course of the infection. The study of seminal fractions will make it possible to monitor the efficiency of sperm preparation methods in obtaining virus-free spermatozoa. In addition to the pathophysiological knowledge that this study will provide, the results will help to define the appropriate course of action and improve the viral safety of medically assisted reproduction in epidemic situations and for patients returning from epidemic areas.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 45 years.
* Patient in the acute phase of CHIKV infection, presenting clinical criteria (known onset of clinical symptoms) that, while not specific, can be highly suggestive in an epidemic area, such as: fever, fatigue, nausea, rash, arthritis/arthralgia, myalgia, headaches, conjunctivitis, and ocular pain.
* Detection of Chikungunya virus genome by Reverse Transcriptase polymerase chain reaction in blood or urine.
* Patient capable of traveling to the laboratory for sample collection.
* Patient who has given informed and voluntary consent and signed the consent form.
* Patient affiliated with a social security system or equivalent.

Exclusion Criteria:

* Patients with an ejaculation disorder, unable to provide a semen sample, or with an abnormal semen volume (<1.5 mL).
* Patient with confirmed male infertility.
* Patients under judicial protection, guardianship, or curatorship.
* Patient already included in another research protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — this study aims to detect the presence of the Chikungunya virus in sperm, so only men can take part.
Enrollment: 15 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Chikungunya virus genomic RNA in sperm | 6 months
  Search for presence of Chikungunya virus genomic RNA in patients sperm when they are in the acute phase of the infection with reverse transcriptase polymerase chain reaction (RT-PCR)

SECONDARY OUTCOMES:
Identification of the exact localization of Chikungunya genomic RNA in semen | 6 months
  polymerase chain reaction based identification of the exact localization of CHIKV genomic RNA, after centrifugation of semen aliquots to separate seminal plasma and seminal cells.
Validation of the efficacy of sperm preparation techniques to isolate Chikungunya-free sperm | 6 months
  Both unprocessed and prepared samples will be tested for the presence of Chikungunya virus RNA using validated real-time reverse transcription PCR (RT-PCR). By comparing the presence of CHIKV RNA before and after sperm preparation, the study aims to determine the capacity of these techniques to produce virus-free sperm. A negative result in the post-preparation sample indicates successful removal of the virus, supporting the potential use of ART in men previously infected with Chikungunya.

CONTACTS AND LOCATIONS:
Overall Officials: Louis BUJAN, Study Chair — University Hospital, Toulouse
Locations (2):
- France (2):
  - CHU de Toulouse, Toulouse, Occitanie
  - CHU Réunion, Saint-Pierre, Réunion

IPD SHARING:
Plan to Share IPD: No